CLINICAL TRIAL: NCT04450901
Title: A Phase 1/2a, Open-Label, Multicenter, Single Arm, Dose Escalation/Dose Expansion Study of YBL-006 in Patients With Advanced Solid Tumors
Brief Title: Dose Escalation/Dose Expansion Study of YBL-006 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Y Biologics Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YBL006C101
Record Dates: First submitted 2020-06-08; First posted 2020-06-30 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort A1 group (Experimental): YBL-006 will be administered once every 2 weeks (Q2W). Dose: 0.5 mg/kg
  Interventions: Drug: YBL-006
- Cohort A2 group (Experimental): YBL-006 will be administered once every 2 weeks (Q2W). Dose: 2 mg/kg
  Interventions: Drug: YBL-006
- Cohort A3 group (Experimental): YBL-006 will be administered once every 2 weeks (Q2W). Dose: 5 mg/kg
  Interventions: Drug: YBL-006
- Cohort A4 group (Experimental): YBL-006 will be administered once every 2 weeks (Q2W). Dose: 10 mg/kg
  Interventions: Drug: YBL-006
- Cohort B1 (Experimental): Tumor type: Advanced Solid tumor (unresectable, locally advanced, or metastatic and have progressed following all standard treatments or are not suitable for standard treatments).
  YBL-006 will be administered once every 2 weeks (Q2W). Dose: 200 mg
  Interventions: Drug: YBL-006
- Cohort B2 (Experimental): Tumor type: Advanced Solid tumor (unresectable, locally advanced, or metastatic and have progressed following all standard treatments or are not suitable for standard treatments).
  YBL-006 will be administered once every 3 weeks (Q3W). Dose: 300 mg
  Interventions: Drug: YBL-006
- Cohort B2 reserve (Experimental): Tumor type: Advanced Solid tumor (unresectable, locally advanced, or metastatic and have progressed following all standard treatments or are not suitable for standard treatments).
  YBL-006 will be administered once every 2 weeks (Q2W). Dose: 300 mg
  Interventions: Drug: YBL-006
- Cohort B3 (Experimental): Tumor type: Metastatic NSCLC (Non-small-cell lung carcinoma), unresectable or metastatic, MSI-H (microsatellite instability-high) or dMMR (Deficient MisMatch Repair), recurrent or metastatic HNSCC (Head and neck squamous cell carcinoma), non-clear cell RCC (renal cell carcinoma), aSCC (anal squamous cell carcinoma), uterine cervical cancer, cSCC (cutaneous squamous cell carcinoma of the skin), uterine endometrial carcinoma, TMB-H (high tumor mutation burden) tumors, epithelial tumor of the penis (squamous cell carcinoma or adenocarcinoma), neuroendocrine tumor (any origin, pancreatic or non-pancreatic), and nasopharyngeal cancer.
  YBL-006 will be administered once every 2 weeks (Q2W). Dose: 200 mg
  Interventions: Drug: YBL-006

INTERVENTIONS:
Drug: YBL-006 — Route of Administration: IV infusion; 0.5 mg/kg Q2W
  Other Names: Cohort A1
  Arms: Cohort A1 group
Drug: YBL-006 — Route of Administration: IV infusion; 2 mg/kg Q2W
  Other Names: Cohort A2
  Arms: Cohort A2 group
Drug: YBL-006 — Route of Administration: IV infusion; 5 mg/kg Q2W
  Other Names: Cohort A3
  Arms: Cohort A3 group
Drug: YBL-006 — Route of Administration: IV infusion; 10 mg/kg Q2W
  Other Names: Cohort A4
  Arms: Cohort A4 group
Drug: YBL-006 — Route of administration : IV infusion, 200 mg Q2W
  Other Names: Cohort B1
  Arms: Cohort B1
Drug: YBL-006 — Route of administration : IV infusion, 300 mg Q3W
  Other Names: Cohort B2
  Arms: Cohort B2
Drug: YBL-006 — Route of administration : IV infusion, 300 mg Q2W
  Other Names: Cohort B2 reserve
  Arms: Cohort B2 reserve
Drug: YBL-006 — Route of administration : IV infusion, 200mg Q2W
  Other Names: Cohort B3
  Arms: Cohort B3

SUMMARY:
This is a Phase 1/2a, open-label, multicenter, dose-escalation/dose-expansion study of YBL-006, in participants with Advanced Solid Tumors. This multicenter study will be conducted in approximately 11-14 participants in the dose escalation phase, and approximately 39-76 participants in dose expansion phase.

DETAILED DESCRIPTION:
Study will consist of three periods:

1. Screening (up to 28 days)
2. Treatment (28-day, 14-day, or 21-day cycles)
3. Follow-up (up to 3 months) The treatment period will consist of 28-day cycles for the dose escalation phase, and 14-day (Cohorts B1, B2 reserve, and B3) or 21-day (Cohort B2) cycles for the dose expansion phase. Each cycle is comprised of two doses of IP administered as an IV infusion on Days 1 and 15 (dose escalation phase) or one dose of IP administered as an IV infusion on Day 1 (dose expansion phase). The treatment duration will be of 1 year in patients who are responding to the treatment.

Dose Escalation:

An accelerated titration design will be utilized for the lowest dose cohort (0.5 mg/kg) in the dose escalation part. Whereas the traditional 3 + 3 design will be utilized for the higher dose cohorts until the proposed starting dose for the Expansion Cohort is determined

Expansion Cohorts:

Up to four tumor-specific expansion cohorts consisting of approximately 39 to 76 participants will evaluate the safety, efficacy, PK, and PD of YBL-006 at the proposed doses of YBL-006"

ELIGIBILITY:
Inclusion Criteria:

1. Written consent on an IRB/ IEC-approved ICF prior to any study-specific evaluation.
2. Male or female aged ≥18 years (or age of legal adult, whichever is older).
3. Life expectancy of at least 3 months.
4. ECOG performance status of 0 to 1.
5. Availability of archival tumour tissue and consent to provide archival tumour for retrospective biomarker analysis, or consent to undergo a fresh tumour biopsy during screening. Participants who do not have an existing (archived) tumour specimen and are unwilling to undergo a biopsy may be enrolled with prior approval from the Sponsor.
6. For participants in dose escalation only: Histologically confirmed solid tumours (except primary CNS tumours) that are unresectable, locally advanced, or metastatic and have progressed following all standard treatments or is not appropriate for standard treatments.
7. Must have at least one measurable lesion based on RECIST Version 1.1. A previously irradiated lesion can be considered a target lesion if the lesion is well defined, measurable and there is objective evidence of interval increase in size.
8. CNS metastasis must be without evidence of progressive neurological symptoms or requires increasing doses of corticosteroids to control the CNS disease for at least 4 weeks. If a participant requires corticosteroids for management of CNS disease, the dose must have been stable with low-dose (same or less than 10 mg/day prednisone or equivalent) for at least two weeks preceding C1D1.
9. Immunosuppressive doses of systemic medications, such as steroids (doses > 10 mg/day prednisone or equivalent) must be discontinued at least 2 weeks before IP administration.
10. Prior surgery that required general anaesthesia must be completed at least 14 days before IP administration. Surgery requiring local/epidural anaesthesia must be completed at least 72 hours before IP administration and participants should be recovered.
11. Adequate haematological and biological function, confirmed by the following laboratory values:

    Neutrophils ≥ 1000/μL Platelets ≥ 75,000/μL Haemoglobin ≥ 9.0 g/dL (may have been transfused) Creatinine ≤ 1.5×upper limit of normal (ULN) Aspartate aminotransferase (AST) ≤ 2.5×ULN (Except with liver metastasis, AST ≤ 5×ULN) Alanine aminotransferase (ALT) ≤ 2.5×ULN (Except with liver metastasis, AST ≤ 5×ULN) Bilirubin ≤ 1.5×ULN (except participants with Gilbert's syndrome, who must have total bilirubin < 3.0 mg/dL).
12. Women must meet 1 of the following criteria: postmenopausal for at least 24 consecutive months; surgically incapable of bearing children (i.e., have had a hysterectomy or bilateral oophorectomy); or utilizing a reliable form of contraception. In general, the decision for appropriate methods to prevent pregnancy should be determined via discussions between the Investigator and the study participant. WOCBP must agree to use a reliable form of contraceptive during the study Treatment Period and for at least 120 days following the last dose of IP.
13. Men must agree to the use of acceptable contraceptive use and avoid sperm donation, during the study Treatment Period and for at least 180 days after the last dose of IP.
14. For the Expansion Cohort, participants enrolling must also meet the following inclusion criteria:

Confirmed diagnosis of one of the following tumour types:

1. For all Expansion Cohorts (B1, B2, B2 reserve, and B3), histologically confirmed advanced solid tumours (except primary CNS tumours) that are unresectable, locally advanced, or metastatic and have progressed following all standard treatments, or are not appropriate for standard treatments.
2. For the B3 cohort, participants must meet one of the following:

   * Participants must have progressed following at least one line of standard systemic therapy and there must not be other approved/standard therapy available that has been shown to prolong overall survival (i.e., in a randomized trial against another standard treatment or by comparison to historical controls); participants who cannot receive other standard therapy that has been shown to prolonged survival due to medical issues will be eligible, if other eligibility criteria are met; OR
   * Participants for whom no standard treatment exists that has been shown to prolong overall survival.

The following tumour types are eligible for the B3 cohort:

- Metastatic NSCLC: Histologically or cytologically confirmed diagnosis of stage IV NSCLC (cases of non-squamous cell carcinoma or NSCLC of unknown subtype) with high (≥ 50%) PD-L1 tumour expression as determined by IHC, without EGFR sensitizing (activating) mutation by PCR and anaplastic lymphoma kinase (ALK) translocation as determined by IHC or fluorescence in situ hybridization (FISH). For pathologically confirmed squamous cell carcinoma, only high (≥ 50%) PD-L1 tumour expression is required.

For Korea only, participants may be enrolled, provided all of the following requirements are met:

* Participants who have failed standard care of anti-cancer treatments, including platinum-based chemotherapy.
* Participants who have refused or discontinued platinum-based chemotherapy due to intolerance.
* Participants who have refused the approved immune checkpoint inhibitors as standard treatment or discontinued due to intolerance. c. Unresectable or metastatic solid tumours with MSI-H or dMMR, locally confirmed by polymerase chain reaction (PCR) or any other appropriate method, such as IHC, in accordance with local site practices:

No additional MSI-H test is required if this test has been completed previously. However, if the participant did not proceed with this test, then additional testing should be completed at a local facility.

d. Histologically confirmed diagnosis of non-clear cell renal cell carcinoma (RCC), anal squamous cell carcinoma (aSCC), uterine cervical cancer, cutaneous squamous cell carcinoma of the skin (cSCC), uterine endometrial carcinoma, tumours which are tumour mutational burden-high (TMB-H), epithelial tumour of the penis (squamous cell carcinoma or adenocarcinoma), neuroendocrine tumour (any origin, pancreatic or non-pancreatic), and nasopharyngeal cancers.

TMB-H: ≥ 10 mutations/megabase, determined at the local (site) laboratory is acceptable for study enrolment.

e. Histologically or cytologically confirmed recurrent or metastatic HNSCC.

Exclusion Criteria:

1. History of severe hypersensitivity reactions to other monoclonal antibodies.
2. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
3. Chemotherapy, radiation therapy, biological cancer therapy, or tyrosine kinase inhibitor (TKI) therapy within 2 weeks or 5 half-lives (whichever is the longer)prior to the first dose of IP, or who has not recovered to National Cancer Institute (NCI)- Common Terminology Criteria for Adverse Events (CTCAE) version 5 or higher Grade 1 or better from the AEs due to cancer therapeutics administered more than 2 weeks earlier; (palliative radiation treatment with a limited field of radiation is allowed up to 14 days prior to first dose of YBL-006).
4. Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast, or localized prostate cancer.
5. Active infection (viral, bacterial, or fungal) requiring IV antimicrobial treatment within 14 days before the first dose of YBL-006.
6. Has known chronic Hepatitis B (e.g., HBsAg reactive) without sufficient anti-viral treatment (prior treatment duration should be more than 3 months), Hepatitis C infection, or human immunodeficiency virus (HIV).
7. Has active or history of interstitial l.ng disease (ILD), or has had a history of pneumonitis that has required oral or IV steroids.
8. Evidence of bleeding diathesis.
9. Any active or suspected autoimmune disease or a documented history of autoimmune disease, or history of a syndrome that required systemic steroids or immunosuppressive medications, except for participants with vitiligo or resolved childhood asthma/atopy.
10. Receipt of live, attenuated vaccine within 28 days prior to the first dose of IP (Note: Participants, if enrolled, should not receive live vaccine during the study and 180 days after the last dose of IP). Vaccination with a killed vaccine is permitted at any time with consultation with the Medical Monitor. Patients may receive vaccination for SARS-CoV-2 (DNA or mRNA vaccine) at the discretion of the Investigator as soon as they are eligible, and a vaccine is available.
11. Known current drug or alcohol abuse.
12. Apparent active or latent tuberculosis infection (purified protein derivative [PPD] test is not required) as indicated by any of the following: PPD recently converted to positive; chest x-ray with definitive evidence of active infectious infiltrate.
13. Presence of any other condition that may increase the risk associated with study participation or may interfere with the interpretation of study results, and, in the opinion of the Investigator, would make the participant inappropriate for entry into the study.
14. Concurrent medical condition requiring the use of immunosuppressive medications or immunosuppressive doses of systemic corticosteroids (doses 10 mg/day prednisone or equivalent). Inhaled or intranasal corticosteroids (with minimal systemic absorption) may be continued if the participant is on a stable dose. Non-absorbed intra-articular steroid injections will be permitted.
15. Use of other investigational therapy within 28 days before IP administration.
16. Non-study related minor surgical procedure (e.g. placement of a central venous access port) ≤ 5 days, or major surgical procedure ≤ 21 days, prior to first dose of IP; in all cases, the participant must be sufficiently recovered and stable before treatment administration.
17. Psychiatric illness or social situation that would preclude study compliance.
18. Participant has clinically significant, uncontrolled, cardiovascular disease including congestive heart failure Grade III or IV according to the New York Heart Association (NYHA) classification; myocardial infarction or unstable angina within the previous 6 months, uncontrolled hypertension, or clinically significant, uncontrolled arrhythmias, including bradyarrhythmias that may cause QT prolongation (e.g., Type II second degree heart block or third degree heart block).
19. Participant has a QT interval corrected using Fridericia's formula (QTcF) > 470 msec. Participant has a history of prolonged QT syndrome or Torsades de pointes. Participant has a familial history of prolonged QT syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability measure through Adverse Events/Serious Adverse Events | Measurements at Baseline till Follow up from 90 days of last dose
  Treatment-related adverse events as assessed by CTCAE v5.0 or higher
Safety and tolerability(Incidence of Treatment-Emergent Adverse Events) measure through Vital Sign- blood pressure | Measurements at Baseline till Follow up from 90 days of last dose
  Measured by result of the Vital Sign- blood pressure
Safety and tolerability(Incidence of Treatment-Emergent Adverse Events) measure through Vital Sign-heart rate | Measurements at Baseline till Follow up from 90 days of last dose
  Measured by result of the Vital Sign- heart rate
Safety and tolerability(Incidence of Treatment-Emergent Adverse Events) measure through 12-lead ECG | Measurements at Baseline till Follow up from 90 days of last dose
  Measured by result of the ECG QT Interval
Safety and tolerability(Incidence of Treatment-Emergent Adverse Events) measure through Physical exam | Measurements at Baseline till Follow up from 90 days of last dose
  Measured by result of the physical exam which includes general appearance, skin, eyes/ears/nose/throat, head and neck.
To establish the recommended Phase 2 dose (RP2D) of YBL-006 in patients with advanced solid tumors | Measurements at Baseline
  Measured through increase in anti-drug antibody (ADA) levels

SECONDARY OUTCOMES:
pharmacokinetic (PK) profile of YBL-006 | Measured at C1D1 till Follow up from 90 days of last dose
  PK is assessed by parameter- area under the curve (AUC)
pharmacokinetic (PK) profile of YBL-006 | Measured at Cycle1(each cycle is 28 days) Day1 till Follow up from 90 days of last dose
  PK is assessed by parameter- maximum (or peak) serum concentration (Cmax)
pharmacokinetic (PK) profile of YBL-006 | Measured at Cycle1(each cycle is 28 days) Day1 till Follow up from 90 days of last dose
  PK is assessed by parameter- time of peak concentration (Tmax)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Jaebong, Study Director — Y-Biologics
Locations (7):
- Macquarie University, Macquarie, New South Wales, Australia
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand